CLINICAL TRIAL: NCT06511414
Title: Effect of Duramesh™ on Hernia Formation After Ileostomy Closure, Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Vitaliy Poylin, Director, Section of Colon and Rectal Surgery, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00220106
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Incisional Hernia; Ileostomy - Stoma
Keywords: duramesh,
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Duramesh (Experimental): using duramesh suture for ileostomy fascial closure
  Interventions: Device: duramesh
- Control (Active Comparator): standard ileostomy fascial closure
  Interventions: Device: Control

INTERVENTIONS:
Device: duramesh — Duramesh™ non-absorbable polypropylene suture is a hollow core, microporous, cylindrical suture made off in polypropylene filaments that are loosely braided and bonded to each other with heat and pressure
  Arms: Duramesh
Device: Control — standard closure of fascia
  Arms: Control

SUMMARY:
Diverting ileostomy is frequently utilized to protect high-risk anastomoses, though it is not shown to reduce the leak rate it may reduce the severe consequences of an anastomotic leak. Ileostomy will be reversed with restoration of continuity in majority of patients. Stoma site incisional hernias after ileostomy closure are complex hernias that can be associated with abdominal pain, discomfort, and a diminished quality of life. Duramesh™ non-absorbable polypropylene suture is a hollow core, microporous, cylindrical suture made off in polypropylene filaments that are loosely braided and bonded to each other with heat and pressure. The Aim of this study is to evaluate Duramesh™ suture vs standard closure on rates of hernia formation after ileostomy closure.

ELIGIBILITY:
Inclusion Criteria:

* • Patients undergoing ileostomy closure after surgery for cancer All patients with a stoma (independent of diagnosis)

  * Age 18 or greater
  * Surgical oncology patient where routine radiologic surveillance for malignancy is planned
  * Patient accepts participation and gives informed consent

Exclusion Criteria:

* • Pregnancy

  * Prior mesh hernia repair at laparotomy site
  * Life expectancy less than 1 years
  * Patient is unable / unwilling to provide informed consent
  * Patient is unable to comply with the protocol or proposed follow-up visits
  * Patient is enrolled in another hernia study
  * Non-English-speaking participants
  * Data from children will not analyzed in this study.
  * Cognitively Impaired Adults: Data from cognitively impaired adults will not analyzed in this study.
  * Adults Unable to Consent: Data from adults unable to consent will not analyzed in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
hernia rates | 1 year
  Compare hernia rates after ileostomy closure between Duramesh™ and standard monofilament closure

SECONDARY OUTCOMES:
infection rate | 1 year
  Evaluate potential side effects including infections and need for re intervention associated with Duramesh™ vs standard closure

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No